CLINICAL TRIAL: NCT02489136
Title: Effect of Spirit Pass on Serum Cortisol Levels, Pain, Physiological Parameters and Haematologic Response in Newborn and Patient
Brief Title: Study of Spirit Pass in Newborn and Patient
Acronym: SSPNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Elida Mara Carneiro da Silva, Elida Mara Carneiro da Silva, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: EMC123
Record Dates: First submitted 2015-05-30; First posted 2015-07-02 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2015-06

CONDITIONS: Pain; Stress
Keywords: spiritist passe; laying of hands; newborn; adult; conditions
MeSH Terms: conditions — Pain; Disease | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spirit Pass (Other): It is a transfusion of psychic energies. Laying of hands to be in front of the incubator or on bed, at a distance at around 10 to 15 cm, during 10 minutes. Evaluate the effects of spirit passe in newborn and adults before and after ten minutes for 3 days.
  Interventions: Other: laying of hands (Spiritist "passe")
- laying of hands by workes (Placebo Comparator): Laying of hand by workers and volunteers, not belonging to Spiritism.Laying of hands to be in front of the incubator or on bed, at a distance at around 10 to 15 cm, during 10 minutes. Evaluate the effects of spirit passe in newborn and adults before and after ten minutes for 3 days.
  Interventions: Other: laying of hands (Spiritist "passe")
- No intervention (No Intervention): No intervention during, in adults before and after ten minutes for 3 days.

INTERVENTIONS:
Other: laying of hands (Spiritist "passe") — In a distance of 10 cm and to apply the spiritist passe for 10 minutes.
  Other Names: laying of hands
  Arms: Spirit Pass; laying of hands by workes

SUMMARY:
Stress is a multiple variable and an inevitable aspect of life. Any change that affects the life of a person is a stressful agent, being possible to widely vary its nature and may be formed by several components, since psychosocial and behavioral factors, such as frustration, anxiety and overload. The goal is to assess the effects of laying on of hands on newborns and patients without direct physical contact. Newborns are allocated in two three groups: G1 - group submitted to imposition of hands by workers, for a period of 10 minutes; G2 group submitted to laying on of hands for 10 minutes; and adults are allocated three groups: G1 - group submitted to imposition of hands by workers, for a period of 10 minutes; G2 group submitted to laying on of hands for 10 minutes; in G3: group without intervention, for a period of 10 minutes.

DETAILED DESCRIPTION:
Individuals responsible for NB will be invited to participate in the research and, after they have signed the informed term of consent, NB will be allocated into two groups (G1 and G2):

G1: group submitted to hand imposition by the workers, for 10 minutes; G2: group submitted to the laying on of hands (spiritist passe), for 10 minutes.

In hospitalized adults, after they have signed the informed term of consent, they will be allocated into three groups:

G1: group submitted to hand imposition by workers and volunteers, not belonging to Spiritism, for 10 minutes; G2: group submitted to the laying on of hands (spiritist passe), for 10 minutes; G3: group with no intervention, for 10 minutes. All interventions will be performed in 3 consecutive days. In group 1 (G1) it will consist of: asking workers and individuals who do not belong to Spiritism to place themselves In front of the incubators or the bed, lay on their hands over the NB or the patient in dorsal decubitus (left hand over the head and the right hand over the chest), in a distance of 10 cm, and emit sincere wishes of improvement to the patient, aiming the healing, for 10 minutes, regardless their belief or religion. Patients will be oriented to direct their thoughts to Jesus during the intervention. For the laying on of hands, Salivary cortisol collection in NB will be carried out in the days: D1 (1st day) and D3 (3rd day). It will be a blind evaluation and allocation of NB and adults in each group. • Anxiety, depression, muscle tension and wellness in adults. [Time Frame: First and third days before and after the interventions.

Diagnosis of each patient included in the study, their beliefs and religions, as well as the characteristics of the passe givers , such as age, gender, time of experience as a passe givers will be analyzed in the characterization of the sample and discussion.

ELIGIBILITY:
Inclusion Criteria:

• It will be included in the study newborns (NB) hospitalized in the nursery and patients aged 18 or over, male and female, conscious and oriented, presenting Glasgow coma scale of 15, hospitalized at the Clinical Hospital of UFTM, who will not be discharged from it for at around the 3 following days.

Exclusion Criteria:

• Individuals who will be excluded from the study:

1. Responsible for the NB or patient who refuses to give the consent, after have been informed;
2. Presence of metabolic diseases, which change the salivary cortisol secretion, verified in their register;
3. NB and adults in mechanical ventilation.

Min Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol | up to third days
  Collection of salivary cortisol will be carried out using wads of cotton. On newborns it will be introduced in the mouth of the baby and left there for at around three minutes and after that, it will be put inside a kit salivette. Cortisol dosage will be by dependent sample.

SECONDARY OUTCOMES:
Anxiety and depression in adults. | First and third days before and after the interventions
  Anxiety and depression in patients will be applied in the questionnaire: Hospital Scale of Anxiety of depression HAD, consisted of 14 items, divided into 7 items of anxiety assessment and 7 of depression.

OTHER OUTCOMES:
Pain | First and third days before and after the interventions
  It will be adopted the Infant Pain Scale (NIPS) in newborns. This scale assesses facial expression, crying, breathing, arms, legs and consciousness. Maximum score is 7 and it is considered pain when all the values are equal or higher than 4.
Physiological parameters | First and third days before and after the interventions
  Physiological parameters such as respiratory frequency, heart frequency and oxygen saturation through Dixtal 2022 monitor in newborn.
Pain | First and third days before and after the interventions
  In adults, it will be adopted the Analogical Visual Scale (AVS), which consists of a horizontal line with 10 centimeters length. In one extremity there is the classification "NO PAIN" and, in the other, "MAXIMUM PAIN".
Physiological parameters | First and third days before and after the interventions
  Physiological parameters such as heart frequency and oxygen saturation through Dixtal 2022 monitor in adults.
Muscle tension in adults. | First and third days before and after the interventions
  Perception of muscle tension in patients will be applied in the questionnaire Analogical scale: analogical visual scale for identification of self-perception of Muscle Tension, individual tension, in which 0 means absence of muscle tension perception and 10 the level of maximum tension perception.
Wellness in adults | First and third days before and after the interventions
  Sense of wellness in patients will be applied in the questionnaire: Analogical scale: analogical visual scale for identification of self-perception of wellness; in which 0 means the absence of wellness perception and 10 the level of maximum wellness perception.

CONTACTS AND LOCATIONS:
Overall Officials: Élida M Carneiro, Mrs., Principal Investigator — Religious and Spiritual Assistance Committee
Locations (1):
- Hospital de Clínicas da UFTM, Uberaba, Minas Gerais, Brazil

REFERENCES:
- [Background] CASTRO M.; MOREIRA A.C. Análise Crítica do Cortisol Salivar na Avaliação do eixo Hipotálamo-Hipófise-Adrenal. Arquivo Brasileiro de Endocrinologia & Metabologia, v. 47, p. 358-367, 2003.
- [Background] Gomes VM, Silva MJ, Araujo EA. [Gradual effects of therapeutic touch in reducing anxiety in university students]. Rev Bras Enferm. 2008 Nov-Dec;61(6):841-6. doi: 10.1590/s0034-71672008000600008. Portuguese. PMID 19142390
- [Background] Selye H. Stress and distress. Compr Ther. 1975 Dec;1(8):9-13. PMID 1222562
- [Background] HOUAISS A.V.; SALLES M. Dicionário Houaiss da Língua. Rio de Janeiro: Editora Objetiva, 2009.
- [Background] LUCCHETTI G. Efeitos do passe espírita no crescimento de culturas de bactérias. Complementary Therapies in Medicine2013;21:627-632.
- [Background] XAVIER F.C. O Consolador. Pelo Espírito Emmanuel. 28. ed. Rio de Janeiro: FEB, 2008.
- [Background] SILVA T.P.; SILVA L.J. Escalas de avaliação da dor utilizadas no recém-nascido. Revisão sistemática. Acta Médica Portuguesa, v. 23, n. 3, p. 437-454, 2010.